CLINICAL TRIAL: NCT06142058
Title: Application of the RecistTM Criteria in Evaluating the Efficacy of Targeted Therapy for Advanced Non-small Cell Lung Cancer With Positive Driving Genes
Brief Title: RecistTM Criteria in Evaluating the Efficacy of Targeted Therapy for NSCLC
Status: Recruiting | Type: Observational
Sponsor: Xueqin Yang (Other)
Responsible Party: Sponsor-Investigator, Xueqin Yang, Prof., Third Military Medical University
Organization: Third Military Medical University (Other)
Other Study IDs: RecistTM-1
Record Dates: First submitted 2023-10-31; First posted 2023-11-21 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Evaluation; NSCLC; Targeted Therapy
Keywords: tumor marker; NSCLC; RECIST; RecistTM; positive driving gene
MeSH Terms: interventions — Response Evaluation Criteria in Solid Tumors

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Patient ctDNA samples are used for NGS detections, with each patient planning to take blood 3-4 times。
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: RecistTM criteria — RecistTM criteria and RECIST criteria were used to evaluate the efficacy of targeted therapy for NSCLC with positive driving gene.
  Other Names: RECIST criteria

SUMMARY:
Investigators established the efficacy evaluation criteria for tumor markers (RecistTM) in the preliminary research. Among patients with advanced non-small cell lung cancer, patients with positive driving genes are more likely to exhibit abnormalities in tumor markers, which suggests that this criteria may be more suitable for evaluating the efficacy of targeted therapy in driving gene positive patients. Moreover, The judgment rules of the prelimary criteria still need further improvement. Therefore, in order to broaden the application scope of the RecistTM criteria, further improve the evaluation rules of RecistTM criteria, and multi-dimensionally confirm the reliability of RecistTM criteria on efficacy evaluation, investigators plan to conduct research on the application of RecistTM criteria in evaluating the efficacy of targeted therapy for advanced non-small cell lung cancer with positive driving genes.

DETAILED DESCRIPTION:
Investigators established the efficacy evaluation criteria for tumor markers (RecistTM) in the preliminary research. The establishment of this criteria makes the application of tumor markers in clinical efficacy evaluation more objective and solves the problem of consistency in clinical efficacy evaluation. Among patients with advanced non-small cell lung cancer, patients with positive driving genes are more likely to exhibit abnormalities in tumor markers, which suggests that this criteria may be more suitable for evaluating the efficacy of targeted therapy in driving gene positive patients. Moreover, The judgment rules of the preliminary criteria still need further improvement. . Therefore, in order to broaden the application scope of the RecistTM criteria, further improve the evaluation rules of RecistTM criteria, and multi-dimensionally confirm the reliability of RecistTM criteria on efficacy evaluation, investigators plan to conduct research on the application of RecistTM criteria in evaluating the efficacy of targeted therapy for advanced non-small cell lung cancer with positive driving genes. Investigators used statistical analysis to assess the consistency of efficacy evaluation between the RecistTM criteria and the RECIST criteria, the correlation between different efficacy and progression free survival (PFS) under the RecistTM, and the correlation between the efficacy of RecistTM criteria and ctDNA level.

ELIGIBILITY:
Inclusion Criteria:

* NSCLC patients with stage IIIB-IV
* Driver gene positive (EGFR,ALK,C-MET, ROS,RET, HER2);
* First line targeted therapy.
* Performance status of 0-2 on the ECOG criteria.
* Any one of the tumor markers is more than three times higher than the normal level, and the tumor markers include: CEA>15ng/ml,CA-199>105U/ml,CA-125>105 U/ml, NSE>60 ng/ml, SCCAg>7.5 ng/ml, CYFRA21-1>21 ng/ml, et al.
* Measurable lesions present
* Age>=18
* Adequate hematologic (neutrophil count >= 1,500/uL, platelets >= 60,000/uL,hemoglobin≥70g/L), hepatic (transaminase =< upper normal limit(UNL)x2.5, bilirubin level =< UNLx1.5), and renal (creatinine =< UNL) function.
* Informed consent from patient or patient's relative.

Exclusion Criteria:

* Patients with dysphagia;
* Unable to taking medication on time;
* Patients with a history of abuse of psychotropic substances who are unable to quit or have mental disorders

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: NSCLC patients with stage IIIB-IV，Driver gene positive， and any one of the tumor markers is more than three times higher than the normal level,
Sampling Method: Non-Probability Sample
Enrollment: 44 (Estimated)
Dates: Start 2023-11-13 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Evaluation consistency | efficacy evaluation at the 1st, 3rd, 6th month after treatment, and every 3 months thereafter up to 1 year
  The ratio of the number of patients with the same efficacy evaluated both by RecistTM and Recist criteria to the total number of the patients.

SECONDARY OUTCOMES:
progression-free survival （PFS） | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 60 months
  The correlation between the efficacy evaluation results of the RecistTM criteria and the RECIST criteria and PFS

OTHER OUTCOMES:
The correlation between the efficacy evaluation results of the RecistTM criteria and the results of ctDNA testing | At the 1st, 3rd, 6th month after treatment, and at the time of disease progression, up to 2 years
  The correlation between the efficacy evaluated by the RecistTM criteria and the ctDNA amounts detected by NGS

CONTACTS AND LOCATIONS:
Locations (1):
- Cancer Center, Dapping Hospital, Army Medical Center of PLA, Chongqing, Chongqing Municipality, China